CLINICAL TRIAL: NCT01136993
Title: Finnish Telestroke Pilot 2007-2009
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Kuusankoski Regional Hospital Kuusankoski Finland (Unknown); Kymenlaakso Central Hospital Kotka Finland (Other); Tampere University Hospital (Other); Central Hospital of Lapland Rovaniemi Finland (Unknown); South Carelia Central Hospital (Other); Länsi-Pohja Central Hospital Kemi Finland (Unknown)
Responsible Party: Dr. Tiina Sairanen, Department of Neurology, HUCH, Helsinki, Finland
Other Study IDs: M1010NL0002
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Stroke
Keywords: Stroke; Thrombolysis; Telestroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All bi-directional telestroke consultations

SUMMARY:
Objective is to describe two years experience from The Finnish Telestroke piloting between Helsinki University Central Hospital (HUCH), Department of Neurology, The Hub, and five hospitals, the spokes. The participating hospitals are from Rovaniemi (Lapland), Kemi (North-West of Finland), Lappeenranta, Kuusankoski and Kotka from South-East of Finland. All the participating hospitals have a stroke unit and the thrombolysis treatment and the follow up of the patients are carried in the treating hospital. The aim of the pilot is to provide these hospitals expertise in thrombolysis treatment during off-hours through teleconsultations.

The teleconsultations were begun between the participating hospitals 05/2007 after about 1 years preparation period. During the preparation period the staff from participating hospitals were trained with simulation training and lectures held by the local staff and the faculty of the Helsinki University hospital.

Telestroke consultation: During two way interactive audio-visual consultation the thrombolysis decision is based on: 1) the consultant going through a check up list of indications and no contraindications to the treatment together with the treating physician and 2) Clinical assessment of NIHSS by the treating physician under guidance of the consultant through the two way video system besides 3) Evaluation of the head CT scan.

The data registered is based on documents made at HUCH and the follow up data provided by the chief neurologist of the other hospitals. 109 teleconsultations have been documented over 2 years period. A unique feature of the Finnish pilot is the high percentage of consultations leading to thrombolysis treatment. Another special feature is that the consultant does the teleconsultation work besides other on call duties.

ELIGIBILITY:
Inclusion Criteria:

* All stroke patients inside 4.5 hours from the symptom onset considered as thrombolysis candidates by the treating physician of the spoke. In suspected basilar artery thrombosis up to 48 h from symptom onset.

Exclusion Criteria:

* Symptom onset > 4.5 h

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All teleconsultations on stroke thrombolysis decision between the Hub (HUCH) and the 5 Spokes during 2 years time period.
Sampling Method: Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of thrombolysis treatments per consultations | 2 years

SECONDARY OUTCOMES:
Safety (sICH) and Efficacy (mRS at 3 months) compared with on-site thrombolysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Sairanen, MD, PhD, Principal Investigator — Department of Neurology, HUCH, Helsinki, Finland
Locations (1):
- Department of neurology, HUCH, Helsinki, Finland

REFERENCES:
- [Background] Tatlisumak T, Soinila S, Kaste M. Telestroke networking offers multiple benefits beyond thrombolysis. Cerebrovasc Dis. 2009;27 Suppl 4:21-7. doi: 10.1159/000213055. Epub 2009 Jun 18. PMID 19546538